CLINICAL TRIAL: NCT00804427
Title: Effect of Fish Oil as an Ethyl Ester or Triglyceride Preparation on Plasma Triglycerides in Hypertriglyceridemic Adults
Brief Title: Effect of Fish Oil on Plasma Triglycerides in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Nordic Naturals (Industry)
Responsible Party: Principal Investigator, Christopher Gardner, Professor of Medicine (Research), Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SU-12042008-1358
Record Dates: First submitted 2008-12-04; First posted 2008-12-08 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Hypertriglyceridemia
Keywords: Fish oil; Triglycerides; Low-density Lipoprotein (LDL) cholesterol; Low-density Lipoprotein (LDL) subclass; Low-density Lipoprotein (LDL) particle size; Low-density Lipoprotein (LDL) phenotype
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Fish Oils; Triglycerides; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fish oil (90% triglycerides) (Experimental): Fish oil (4 grams/day of combined EPA and DHA) as 90% triglyceride formulation, taken in two divided doses with main meals.
  Interventions: Dietary Supplement: Fish oil (90% triglycerides)
- Fish oil (60% triglycerides) (Experimental): Fish oil (4 grams/day of combined EPA and DHA) as 60% triglyceride formulation, taken in two divided doses with main meals.
  Interventions: Dietary Supplement: Fish oil (60% triglycerides)
- Fish oil (ethyl esters) (Experimental): Fish oil (4 grams/day of combined EPA and DHA) as ethyl esters formulation (0% triglycerides), taken in two divided doses with main meals.
  Interventions: Dietary Supplement: Fish oil (ethyl esters)
- Soy oil (Placebo Comparator): Soy oil supplement with identical total fat content, taken in two divided doses with main meals.
  Interventions: Dietary Supplement: Soy oil

INTERVENTIONS:
Dietary Supplement: Fish oil (90% triglycerides)
  Arms: Fish oil (90% triglycerides)
Dietary Supplement: Fish oil (60% triglycerides)
  Arms: Fish oil (60% triglycerides)
Dietary Supplement: Fish oil (ethyl esters)
  Arms: Fish oil (ethyl esters)
Dietary Supplement: Soy oil
  Arms: Soy oil

SUMMARY:
The purpose of this small, short pilot study is to determine the feasibility (e.g., recruitment, dose acceptance, retention) of a future longer trial comparing the effects of two types of omega-3 fats from fish oil on plasma triglycerides. The two types of fish oil are composed of (1) omega-3 fatty acids in triglyceride form; and (2) as esterified free fatty acids (i.e. ethyl esters). Although these two types of fish oil supplements are available to the public, it remains unclear whether they are equally effective in lowering plasma triglycerides.

DETAILED DESCRIPTION:
This study is a double-blinded, parallel design, placebo controlled trial with three active treatment arms to compare the triglyceride (TG) lowering effects of the same dose of EPA and DHA provided in three formulations of supplements that differ in the proportion of omega-3 FA present as ethyl esters vs. triglycerides. The active therapy for each of the three fish oil supplementation arms is 4 g/day of combined EPA and DHA provided as: a) 90% TG formulation, b) 60% TG formulation, or c) ethyl esters (esterified fatty acids)(i.e., 0% TG). The placebo was a soy oil supplement with an identical total fat content. The primary outcome is the 12-week change in TG concentrations in the active groups vs. placebo. Secondary outcomes include LDL particle distribution, defined as either subclasses LDL1, LDL2, LDL3 and LDL4, and LDL subclass phenotype patterns A, B, or A/B.

ELIGIBILITY:
Inclusion Criteria:*Gender: Both women and men

* Age: > or = 18 years
* Ethnicity and race: All ethnic and racial backgrounds welcome
* Fasting blood triglycerides greater than or equal to 150 mg/dL
* Planning to be available for clinic visits for the 12 weeks of study participation
* Ability and willingness to give written informed consent
* No known active psychiatric illness. Exclusion Criteria:*At screening:
* Daily intake of dietary supplements containing omega-3 FAs within the past month.
* Fasting blood glucose greater than or equal to 126 mg/dL
* Self reported personal history of:
* Clinically significant atherosclerosis (e.g., CAD, PAD)
* Malignant neoplasm
* Subjects currently receiving the following medications (self report):
* Lipid lowering drugs including statins
* Anti-hypertensive drugs: beta-blockers and thiazides
* Body Mass Index (BMI) greater than or equal to 40.
* Pregnant or Lactating
* Inability to communicate effectively with study personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-12; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Triglycerides at 3 months | Baseline and 3 months
  Change was calculated as the value at 3 months minus the value at baseline

SECONDARY OUTCOMES:
Change from baseline in LDL particle concentration (LDL1, LDL2, LDL3, LDL4) at 3 months | Baseline and 3 months
  Change was calculated as the value at 3 months minus the value at baseline
Change from baseline in LDL phenotype pattern (A, B, or A/B) at 3 months | Baseline and 3 months
  Change was calculated as the number (and percent) of participants who improved their LDL phenotype pattern at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Gardner, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oelrich B, Dewell A, Gardner CD. Effect of fish oil supplementation on serum triglycerides, LDL cholesterol and LDL subfractions in hypertriglyceridemic adults. Nutr Metab Cardiovasc Dis. 2013 Apr;23(4):350-7. doi: 10.1016/j.numecd.2011.06.003. Epub 2011 Sep 15. PMID 21924882
- See also: Description of study and summary of results — https://med.stanford.edu/nutrition/research/completed-studies/fish-oil-and-triglycerides.html